CLINICAL TRIAL: NCT05081388
Title: A Phase 1/2/3 Adaptive Study to Evaluate the Safety, Tolerability, and Efficacy of REGN14256+Imdevimab for the Treatment of COVID-19 Patients Without Risk Factors for Progression to Severe Disease
Brief Title: COVID-19 Study to Evaluate Safety, Tolerability, and Efficacy of REGN14256+Imdevimab for the Treatment of COVID-19 Adult and Adolescent Patients Without Risk Factors for Progression to Severe Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R14256-COV-2149
Record Dates: First submitted 2021-10-14; First posted 2021-10-18 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: SARS-CoV-2
Keywords: COVID-19; Non-hospitalized; Low-risk; Symptomatic; Coronavirus disease 2019 (COVID-19); Severe acute respiratory syndrome coronavirus 2 (SARS-COV-2); coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — REGN14256; imdevimab; casirivimab and imdevimab drug combination; casirivimab

STUDY DESIGN:
Intervention Model Description: Phase1/Phase2/Phase3
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- REGN14256 + imdevimab (Experimental): Phase 1, Phase 2: Randomized 1:1:1:1:1 Phase 3: (≥18 Years): Randomized 1:1:1 Phase 3: (Open label) (≥12 and <18 Years)
  Interventions: Drug: REGN14256; Drug: imdevimab
- REGN14256 (Experimental): Phase 1, Phase 2: Randomized 1:1:1:1:1
  Interventions: Drug: REGN14256
- Imdevimab (Experimental): Phase 1, Phase 2: Randomized 1:1:1:1:1
  Interventions: Drug: imdevimab
- casirivimab + imdevimab (Experimental): Phase 1, Phase 2: Randomized 1:1:1:1:1 Phase 3: (≥18 Years): Randomized 1:1:1
  Interventions: Drug: imdevimab; Drug: casirivimab + imdevimab
- Placebo (Experimental): Phase 1, Phase 2: Randomized 1:1:1:1:1 Phase 3: (≥18 Years): Randomized 1:1:1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REGN14256 — Sub-cutaneous (SC) single dose
  Arms: REGN14256; REGN14256 + imdevimab
Drug: imdevimab — SC single dose
  Other Names: REGN10987
  Arms: Imdevimab; REGN14256 + imdevimab; casirivimab + imdevimab
Drug: casirivimab + imdevimab — SC single dose
  Other Names: REGN10933 + REGN10987; REGN-COV2; REGEN-COV™; Ronapreve™
  Arms: casirivimab + imdevimab
Drug: Placebo — SC single dose
  Arms: Placebo

SUMMARY:
Primary Objectives Phase 1 (Safety and Tolerability)

• Evaluate the safety and tolerability of REGN14256+imdevimab and REGN14256 monotherapy, as measured by treatment-emergent adverse events (TEAEs), injection-site reactions (ISRs), and hypersensitivity reactions

Phase 1/2 (Virologic Efficacy) • Evaluate the virologic efficacy of REGN14256+imdevimab and REGN14256 monotherapy compared to placebo, as measured by time-weighted average (TWA) change from baseline in viral load through day 7

Phase 1/2/3 (Clinical Efficacy)

• Evaluate the clinical efficacy of REGN14256+imdevimab compared to placebo, as measured by COVID-19 symptoms resolution

Secondary Objectives Phase 1 (Safety and Tolerability) • Evaluate the safety and tolerability of REGN14256+imdevimab and REGN14256 monotherapy, as measured by treatment-emergent serious adverse events (SAEs)

Phase 2 and Phase 3 (Safety and Tolerability)

• Evaluate the safety and tolerability of REGN14256+imdevimab and REGN14256 monotherapy, as measured by TEAEs, ISRs, hypersensitivity reactions, and SAEs

Phase 1, Phase 2, and Phase 3 (Virologic Efficacy, Drug Concentration, and Immunogenicity)

* Evaluate additional indicators of virologic efficacy of REGN14256+imdevimab and REGN14256 monotherapy
* Characterize the concentration-time profile of REGN14256 administered in combination with imdevimab or alone as a monotherapy
* Assess the immunogenicity of REGN14256 administered in combination with imdevimab or alone as a monotherapy

ELIGIBILITY:
Phase 1 will enroll adult patients (≥18 years of age), Phase 2 will enroll adult patients, Phase 3 will enroll adult patients and an additional adolescent cohort of patients (≥12 and <18 years of age)

Key Inclusion Criteria:

1. For the adolescent cohort in Phase 3 only: Weighs ≥40 kg at randomization
2. Has SARS-CoV-2-positive antigen or molecular diagnostic test (by validated SARSCoV-2 antigen, RT-PCR, or other molecular diagnostic assay, using an appropriate sample such as nasopharyngeal [NP], nasal, oropharyngeal [OP], or saliva) ≤72 hours prior to randomization. A historical record of a positive result is acceptable as long as the sample was collected ≤72 hours prior to randomization
3. Has symptoms consistent with COVID-19 (as determined by the investigator) with onset ≤7 days before randomization, and doesn't have a medical condition or other factors associated with high risk for progression to severe COVID-19 as outlined in the exclusion criteria
4. Maintains O2 saturation ≥93% on room air

Key Exclusion Criteria:

1. Has a medical condition or other factors associated with high risk for progression to severe COVID-19:

   1. Cancer
   2. Cardiovascular disease (such as heart failure, coronary artery disease, cardiomyopathies, congenital heart disease or hypertension)
   3. Chronic lung disease including chronic obstructive pulmonary disease, asthma (moderate to severe), interstitial lung disease, cystic fibrosis, and pulmonary hypertension
   4. Chronic kidney disease at any stage
   5. Chronic liver disease (such as alcohol-related, nonalcoholic fatty liver disease, cirrhosis)
   6. Dementia or other chronic neurological condition
   7. Diabetes mellitus (type 1 or type 2)
   8. Immunodeficiency disease or taking immunosuppressive treatment
   9. Medical-related technological dependence [for example, tracheostomy, gastrostomy, or positive pressure ventilation (not related to COVID-19)]
   10. Neurodevelopmental disorder (for example, cerebral palsy) or other condition that confers medical complexity (for example, genetic or metabolic syndromes and severe congenital anomalies)
   11. Overweight (defined as BMI >25 kg/m2) or obesity (defined as BMI ≥30 kg/m2)
   12. Poorly controlled HIV infection or AIDS
   13. Pregnancy
   14. Sickle cell disease or thalassemia
   15. Stroke or cerebrovascular disease
2. Prior, current (at randomization) or planned use (within time period given per CDC guidance [90 days]) of any authorized or approved vaccine for COVID-19
3. Was admitted to a hospital for COVID-19 prior to randomization, or is hospitalized (inpatient) for any reason at randomization
4. Has a known prior SARS-CoV-2 infection or positive SARS-CoV-2 serologic test
5. Has a positive SARS-CoV-2 antigen or molecular diagnostic test from a sample collected >72 hours prior to randomization
6. Has participated, or is participating, in a clinical research study evaluating COVID-19 convalescent plasma, mAbs against SARS-CoV-2, or intravenous immunoglobulin (IVIG) within 3 months or within 5 half-lives of the investigational product (whichever is longer) prior to the screening visit
7. Prior, current, or any of the following treatments: COVID-19 convalescent plasma, mAbs against SARS-CoV-2, IVIG (any indication), systemic corticosteroids (any indication), or COVID-19 treatments (authorized, approved, or investigational)
8. Has known active infection with influenza or other non-SARS-CoV-2 respiratory pathogen, confirmed by a diagnostic test
9. Has been discharged, or is planned to be discharged, to a quarantine center
10. Has participated, is participating, or plans to participate in a clinical research study evaluating any authorized, approved, or investigational vaccine for COVID-19
11. For Phase 1only: Women of childbearing potential (WOCBP) who are unwilling to practice highly effective contraception prior to the initial dose/start of the first treatment and for at least 6 months after study drug administration as described in the protocol

Note: Other protocol-defined inclusion/ exclusion criteria apply

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (27):
- United States (27):
  - Regeneron Research Site, La Mesa, California
  - Ark Clinical Research, Long Beach, California
  - PNS Clinical Research, LLC, Mission Viejo, California
  - Regeneron Research Site, Ft. Pierce, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Regeneron Research Site, Loxahatchee Groves, Florida
  - Project 4 Research, Inc., Miami, Florida
  - Universal Medical and Research Center, LLC, Miami, Florida
  - Global Medical Trials, Miami, Florida
  - Bio-Medical Research LLC, Miami, Florida
  - Charisma Research and Medical Center, Miami Lakes, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Regeneron Research Site, Winter Park, Florida
  - IACT Health, Columbus, Georgia
  - Chicago Clinical Research Institute, Chicago, Illinois
  - Regeneron Research Site, Ames, Iowa
  - Regeneron Research Site, Marrero, Louisiana
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Forte Family Practice, Las Vegas, Nevada
  - New York Health and Hospitals / Lincoln, The Bronx, New York
  - NYC H+H / Jacobi Medical Center, The Bronx, New York
  - Regeneron Research Site, Wilmington, North Carolina
  - Regeneron Research Site, Dayton, Ohio
  - Carolina Medical Research, Clinton, South Carolina
  - PharmaTex Research, LLC, Amarillo, Texas
  - Advanced Diagnostics Clinic, River Oaks Hospital and Clinics, Houston, Texas
  - Regeneron Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was initiated in November 2021, however, due to the reduced activity of REGN14256+imdevimab against the emerging Omicron variant and not due to any safety concerns, study enrollment was paused and later terminated. As a result, only 25 participants were randomized into the phase 1 portion of the study and the phase 2 and phase 3 portions of the study were never opened.
Pre-assignment Details: The study was initiated in November 2021, however, due to the reduced activity of REGN14256+imdevimab against the emerging Omicron variant and not due to any safety concerns, study enrollment was paused and later terminated. As a result, only 25 participants were randomized into the phase 1 portion of the study and the phase 2 and phase 3 portions of the study were never opened
Groups:
- Placebo; Imdevimab (600 mg SC); REGN14256 (600 mg SC); Casirivimab + Imdevimab (1200 mg SC); REGN14256 + Imdevimab (1200 mg SC): Phase 1 only. Phase 2 and Phase 3 portions of the study were never opened
Period: Overall Study
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Started | 4 | 5 | 6 | 6 | 4
Completed | 3 | 4 | 6 | 5 | 4
Not Completed | 1 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Subject decision | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC) | Total
Number analyzed (Participants) | 4 | 5 | 6 | 6 | 4 | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.8 (1.50) | 50.4 (14.05) | 38.2 (19.81) | 30.3 (7.87) | 42.0 (9.90) | 37.4 (14.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 3 | 2 | 11
  Male | 2 | 3 | 4 | 3 | 2 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 3 | 6 | 3 | 19
  Not Hispanic or Latino | 1 | 1 | 3 | 0 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 0 | 3
  White | 3 | 5 | 5 | 5 | 4 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events (TEAEs)
Description: Phase 1
Time Frame: Through Day 29
Population: The study was terminated in the Phase 1 portion of the study. The Safety Analysis Set (SAF) includes all randomized participants who received any study drug; it is based on the treatment received. Only Phase 1 data was collected. Phase 2 and Phase 3 portions of the study were never opened.
Measure: Number; unit: Events
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 4
Events | 1 | 3 | 1 | 1 | 2

2. Primary Outcome: Severity of TEAEs
Description: Severity was based on Grading. Grade 1 was less severe. Grade 5 was more severe.
  1. - Mild; Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
  2. - Moderate; Minimal, local, or noninvasive intervention indicated; limiting age appropriate instrumental activities of daily living (ADL)
  3. - Severe; Severe or medically significant but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; disabling; ADL2 limiting self-care
  4. - Life-threatening; Life threatening consequences; urgent intervention indicated
  5. - Death; Death related to adverse events
Time Frame: Through Day 29
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 4
Participants
  With at least one Grade 1 TEAE | 0 | 2 | 1 | 1 | 2
  With at least one Grade 2 TEAE | 1 | 0 | 0 | 0 | 0
  With at least one Grade 3 TEAE | 0 | 1 | 0 | 0 | 0
  With at least one Grade 4 TEAE | 0 | 0 | 0 | 0 | 0
  With at least one Grade 5 TEAE | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Injection-site Reactions (ISRs)
Description: Phase 1 only
Time Frame: Through Day 169
Population: The Safety Analysis Set (SAF) includes all randomized participants who received any study drug; it is based on the treatment received. The study was terminated during Phase 1. Only Phase 1 data was collected. Phase 2 and Phase 3 portions of the study were never opened.
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 4
Percentage of Participants | 0 | 0 | 0 | 0 | 25.0

4. Primary Outcome: Severity of ISRs (Injection Site Reactions)
Description: Severity was based on Grading. Grade 1 was less severe. Grade 5 was more severe.
  Grade 1 - Tenderness with or without associated symptoms (eg, warmth, erythema, itching) Grade 2 - Pain; lipodystrophy; edema; phlebitis Grade 3 - Ulceration or necrosis; severe tissue damage; operative intervention indicated Grade 4 - Life-threatening consequences; urgent intervention indicated Grade 5 - Death
Time Frame: Through Day 29
Population: as for outcome 3
Measure: Number; unit: Events
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 4
Events
  With at least one Grade 1 ISR | 0 | 0 | 0 | 0 | 1
  With at least one Grade 2 ISR | 0 | 0 | 0 | 0 | 0
  With at least one Grade 3 ISR | 0 | 0 | 0 | 0 | 0
  With at least one Grade 4 ISR | 0 | 0 | 0 | 0 | 0
  With at least one Grade 5 ISR | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Percentage of Participants With Hypersensitivity Reactions
Description: Phase 1
Time Frame: Through Day 169
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 4
Percentage of Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Severity of Hypersensitivity Reactions Over Time
Description: Grade 1 - Systemic intervention not indicated. Grade 2 - Oral intervention indicated Grade 3 - Bronchospasm; hospitalization indicated for clinical sequelae; intravenous intervention indicated Grade 4 - Life-threatening consequences; urgent intervention indicated Grade 5 - Death
Time Frame: Through Day 169
Population: The study was terminated in the Phase 1 portion of the study. The Safety Analysis Set (SAF) includes all randomized participants who received any study drug; it is based on the treatment received. Phase 2 and Phase 3 portions of the study were never opened.
Measure: Number; unit: Events
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 4
Events
  With at least one Grade 1 | 0 | 0 | 0 | 0 | 0
  With at least one Grade 2 | 0 | 0 | 0 | 0 | 0
  With at least one Grade 3 | 0 | 0 | 0 | 0 | 0
  With at least one Grade 4 | 0 | 0 | 0 | 0 | 0
  With at least one Grade 5 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Time-weighted Average (TWA) Daily Change From Baseline in Viral Load (log10 Copies/mL)
Description: Phase 1 Measured by SARS-CoV-2 quantitative reverse transcription polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples
Time Frame: Day 1 to day 7
Population: The modified full analysis set (mFAS) includes all randomized patients with a positive central lab determined SARS-CoV-2 RT-qPCR result from nasopharyngeal (NP) swab samples at randomization and is based on the treatment received. The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened.
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 4 | 6 | 6 | 2
log10 copies/mL | -4.02 (1.461) | -2.28 (0.286) | -2.30 (0.964) | -2.72 (1.517) | -1.76 (0.003)

8. Secondary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: Phase 1
Time Frame: Through Day 169
Population: The Safety Analysis Set (SAF) includes all randomized participants who received any study drug; it is based on the treatment received. The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened.
Measure: Number; unit: Percentage
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 4
Percentage | 33.3 | 20.0 | 0 | 0 | 0

9. Secondary Outcome: TEAEs (Treatment-Emergent Adverse Events)
Description: Phase 2 and Phase 3
Time Frame: Through Day 29
Population: The Safety Analysis Set (SAF) includes all randomized participants who received any study drug; it is based on the treatment received. The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened. No data collected.
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Severity of TEAEs (Treatment-Emergent Adverse Event)
Description: Phase 2 and Phase 3
Time Frame: Through Day 29
Population: as for outcome 9
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With ISRs (Injection-Site Reactions)
Description: Phase 2 and Phase 3
Time Frame: Through Day 169
Population: as for outcome 9
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Severity of ISRs (Injection-Site Reactions)
Description: Phase 2 and Phase 3
Time Frame: Through Day 169
Population: as for outcome 9
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With Hypersensitivity Reactions
Description: Phase 2 and Phase 3
Time Frame: Through Day 169
Population: as for outcome 9
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Severity of Hypersensitivity Reactions Over Time
Description: Phase 2 and Phase 3
Time Frame: Through Day 169
Population: as for outcome 9
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Percentage of Participants With Treatment-emergent SAEs (Serious Adverse Events)
Description: Phase 2 and Phase 3
Time Frame: Through Day 169
Population: The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Time-weighted Average Change From Baseline in Viral Load
Description: Phase 2 and Phase 3
  Time-weighted average (TWA) daily change from baseline in viral load (log10 copies/mL) as measured by SARS-CoV-2 quantitative reverse transcription polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Through Day 169
Population: The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened. No data collected.
Groups:
- Placebo; Imdevimab (600 mg SC); REGN14256 (600 mg SC); Casirivimab + Imdevimab (1200 mg SC): Phase 2 and Phase 3 portions of the study were never opened
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in Viral Load (Phase 1)
Description: Phase 1 Change from baseline in viral load (log10 copies/mL) as measured by SARS-CoV-2 quantitative reverse transcription polymerase chain reaction (RT-qPCR) in nasopharyngeal (NP) swab samples.
Time Frame: Through Day 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 3 | 5 | 6 | 6 | 2
log10 copies/mL
  Change from Baseline to Day 3: number analyzed (Participants) | 3 | 5 | 6 | 6 | 1
  Change from Baseline to Day 3 | -3.93 (2.691) | -2.14 (0.251) | -1.60 (1.598) | -2.27 (1.097) | 0.23 (NA) — Too small a number of data points calculate
  Change from Baseline to Day 5: number analyzed (Participants) | 3 | 5 | 6 | 6 | 1
  Change from Baseline to Day 5 | -5.25 (1.400) | -3.74 (1.585) | -3.28 (1.085) | -3.73 (2.677) | -1.88 (NA) — Too small a number of data points calculate
  Change from Baseline to Day 7: number analyzed (Participants) | 3 | 4 | 6 | 6 | 2
  Change from Baseline to Day 7 | -5.76 (2.220) | -3.02 (1.115) | -4.01 (2.000) | -4.31 (2.121) | -5.37 (2.617)

18. Secondary Outcome: Change From Baseline in Viral Load
Description: Phase 2, and Phase 3 As measured by RT-qPCR in NP samples
Time Frame: Through Day 7
Population: The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened. No data collected.
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Viral Loads Below the Limit of Detection
Description: Phase 1, Phase 2, and Phase 3
Time Frame: Through Day 169
Population: The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened. No data collected.
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Concentrations of REGN14256 in Serum Over Time (Phase 1)
Description: Phase 1
Time Frame: Through Day 169
Population: The PK analysis set includes all treated participants who received REGN14256 and who had at least 1 non-missing result of respective analyte following the first dose of REGN14256. The study was terminated, data was not collected for Phase 2 and Phase 3, as these portions were never opened.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- REGN14256 600 mg SC; REGN14256+Imdevimab (1200 mg SC): Phase 1 only. Phase 2 and Phase 3 portions of the study were never opened
Arm/Group | REGN14256 600 mg SC | REGN14256+Imdevimab (1200 mg SC)
Number analyzed (Participants) | 6 | 4
mg/L
  Pre-dose | 0 (0) | 0 (0)
  Post-dose: number analyzed (Participants) | 6 | 3
  Post-dose | 3.45 (4.36) | 9.66 (10.6)
  Day 1: number analyzed (Participants) | 6 | 3
  Day 1 | 21.5 (16.6) | 52.4 (43.3)
  Day 2: number analyzed (Participants) | 6 | 3
  Day 2 | 37.5 (25.4) | 58.5 (38.3)
  Day 6 | 53.2 (29.9) | 63.6 (26.2)
  Day 28 | 30.7 (15.7) | 39.9 (14.6)
  Day 59: number analyzed (Participants) | 6 | 3
  Day 59 | 13.5 (7.57) | 19.6 (5.78)
  Day 89: number analyzed (Participants) | 6 | 3
  Day 89 | 7.30 (4.46) | 9.03 (3.43)
  Day 119: number analyzed (Participants) | 6 | 3
  Day 119 | 3.44 (2.42) | 4.23 (1.73)

21. Secondary Outcome: Concentrations of REGN14256 in Serum Over Time
Description: Phase 2 and Phase 3
Time Frame: Through Day 169
Population: The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened. No data collected.
Arm/Group | REGN14256 (600 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Concentrations of Imdevimab in Serum Over Time (Phase 1)
Description: Phase 1
Time Frame: Through Day 169
Population: The PK analysis set includes all treated participants who received imdevimab and who had at least 1 non-missing result of respective analyte following the first dose of imdevimab. The study was terminated, data was not collected for Phase 2 and Phase 3, as these portions were never opened.
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Imdevimab 600 mg SC; Casirivimab+Imdevimab (1200 mg SC); REGN14256+Imdevimab (1200 mg SC): Phase 1 only. Phase 2 and Phase 3 portions of the study were never opened
Arm/Group | Imdevimab 600 mg SC | Casirivimab+Imdevimab (1200 mg SC) | REGN14256+Imdevimab (1200 mg SC)
Number analyzed (Participants) | 5 | 6 | 4
mg/L
  Pre-dose | 2.46 (3.59) | 0.398 (0.976) | 0.360 (0.720)
  Post-dose: number analyzed (Participants) | 5 | 6 | 3
  Post-dose | 3.43 (3.13) | 3.06 (2.36) | 9.03 (6.47)
  Day 1: number analyzed (Participants) | 5 | 6 | 3
  Day 1 | 19.7 (9.74) | 31.2 (10.5) | 27.9 (21.0)
  Day 2: number analyzed (Participants) | 5 | 6 | 3
  Day 2 | 28.4 (6.08) | 40.7 (11.8) | 31.9 (19.2)
  Day 6: number analyzed (Participants) | 4 | 5 | 4
  Day 6 | 42.7 (16.8) | 52.2 (16.3) | 38.8 (7.59)
  Day 28: number analyzed (Participants) | 4 | 6 | 4
  Day 28 | 18.9 (9.94) | 27.9 (8.34) | 20.8 (12.2)
  Day 59: number analyzed (Participants) | 4 | 6 | 3
  Day 59 | 7.66 (3.68) | 10.3 (4.40) | 7.18 (3.75)
  Day 89: number analyzed (Participants) | 4 | 5 | 3
  Day 89 | 3.26 (1.80) | 4.37 (2.12) | 3.73 (2.46)
  Day 119: number analyzed (Participants) | 4 | 4 | 3
  Day 119 | 1.72 (1.06) | 2.60 (1.52) | 2.68 (0.910)

23. Secondary Outcome: Concentrations of Imdevimab in Serum Over Time
Description: Phase 2 and Phase 3
Time Frame: Through Day 169
Population: The study was terminated, and Phase 2 and Phase 3 portions of the study were never opened. No data collected.
Arm/Group | Placebo | REGN14256 + Imdevimab (1200 mg SC) | REGN14256 (600 mg SC) | Imdevimab (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Incidence and Titer of Anti-drug Antibodies (ADA) to REGN14256 Over Time
Description: Phase 1, Phase 2, and Phase 3
Time Frame: Through Day 169
Population: As prespecified within the SAP (statistical analysis plan), ADA sample analysis was not performed due to early study termination; therefore, ADA analysis data was not generated. No data collected.
Groups:
- Placebo: Placebo
- Imdevimab (600 mg SC): Imdevimab 600 mg administered subcutaneously
- REGN14256 (600 mg SC): REGN14256 600 mg administered subcutaneously
- Casirivimab + Imdevimab (1200 mg SC): Casirivimab + Imdevimab 1200 mg administered subcutaneously
- REGN14256 + Imdevimab (1200 mg SC): REGN14256 + Imdevimab 1200 mg administered subcutaneously
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Incidence and Titer of ADA to Imdevimab Over Time
Description: Phase 1, Phase 2, and Phase 3
Time Frame: Through Day 169
Population: as for outcome 24
Groups:
- Imdevimab (600 mg SC): Imdevimab (600 mg SC)
- REGN14256 (600 mg SC): REGN14256 (600 mg SC)
- Casirivimab + Imdevimab (1200 mg SC): Casirivimab + Imdevimab (1200 mg SC)
- REGN14256 + Imdevimab (1200 mg SC): REGN14256 + Imdevimab (1200 mg SC)
Arm/Group | Placebo | Imdevimab (600 mg SC) | REGN14256 (600 mg SC) | Casirivimab + Imdevimab (1200 mg SC) | REGN14256 + Imdevimab (1200 mg SC)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to end of study (Up to 169 days)
Groups:
- REGN14256+Imdevimab 1200 mg SC; Casirivimab+Imdevimab 1200 mg SC: Phase 1 only. Phase 2 and Phase 3 portions of the study were never opened
Arm/Group | Placebo | Imdevimab 600 mg SC | REGN14256 600 mg SC | REGN14256+Imdevimab 1200 mg SC | Casirivimab+Imdevimab 1200 mg SC
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/6 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5 | 0/6 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 2/5 | 1/6 | 2/4 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | Imdevimab 600 mg SC (N=5) | REGN14256 600 mg SC (N=6) | REGN14256+Imdevimab 1200 mg SC (N=4) | Casirivimab+Imdevimab 1200 mg SC (N=6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | Imdevimab 600 mg SC (N=5) | REGN14256 600 mg SC (N=6) | REGN14256+Imdevimab 1200 mg SC (N=4) | Casirivimab+Imdevimab 1200 mg SC (N=6)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the reduced activity of REGN14256+Imdevimab against the emerging Omicron variant and not due to any safety concerns, study enrollment was paused and later terminated in the phase 1 portion of the study. Phase 2 and phase 3 portions of the study were never opened. As a result, and due to small sample size, not all of the original objectives and endpoints were analyzed as planned

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT05081388/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/88/NCT05081388/SAP_001.pdf